CLINICAL TRIAL: NCT03208894
Title: Role of Salbutamol and Furosemide in Transient Tachypnea of Newborn
Brief Title: Role of Salbutamol and Furosemide in TTN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Armed Forces Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, arshad khushdil, CONCULTANT PEDIATRICIAN, Armed Forces Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TTN
Record Dates: First submitted 2017-07-01; First posted 2017-07-06 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Transient Tachypnea of the Newborn
MeSH Terms: conditions — Transient Tachypnea of the Newborn | interventions — Furosemide

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- with salbutamol (Experimental)
  Interventions: Drug: Furosemide Injection
- with furosemide (Experimental)
  Interventions: Drug: Furosemide Injection
- both furosemide and salbutamol (Experimental)
  Interventions: Drug: Furosemide Injection
- no inervention (No Intervention)

INTERVENTIONS:
Drug: Furosemide Injection — efficacy of salbutamol and furosemide in TTN
  Other Names: salbutamol inhalation
  Arms: both furosemide and salbutamol; with furosemide; with salbutamol

SUMMARY:
to see the effects of slabutamol and IV furosemide in the treatment of transient tachypnea of newborn

ELIGIBILITY:
Inclusion Criteria:

* all newborn babies with clinically diagnosed TTN

Exclusion Criteria:

* babies less than 34 weeks babies with congenital malformations and CHD

Ages: 1 Hour to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
duration of oxygen requiremment in neonates having TTN. | upto 6 months
  neonates will be subjected to treatment with furosemide and sabutamol and the duration of oxygen dependecy will be assessed.

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - Department of Pediatrics, Rawalpindi, Punjab Province
  - Military Hospital, Rawalpindi, Punjab Province

IPD SHARING:
Plan to Share IPD: No